CLINICAL TRIAL: NCT02971943
Title: Classification of Ankle Injury Observed With X-ray Combined With Magnetic Resonance Imaging: a Retrospective, Self-controlled, Clinical Trial With 3-month Follow-up
Brief Title: Classification of Ankle Injury Observed With X-ray Combined With Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Guobin Liu, Chief Physician, The First Hospital of Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstHebei_001
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Ankle Injury
MeSH Terms: conditions — Ankle Injuries | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- internal fixation for ankle fractures (Other): The patients with ankle injury underwent internal fixation for ankle fractures and ligament repair. Ankle was observed with X-ray and magnetic resonance imaging preoperatively and 3 months postoperatively.
  Interventions: Procedure: internal fixation for ankle fractures

INTERVENTIONS:
Procedure: internal fixation for ankle fractures — The patients with ankle injury underwent internal fixation for ankle fractures and ligament repair. Ankle was observed with X-ray and magnetic resonance imaging.

SUMMARY:
To verify whether X-ray combined with MRI is able to carry out correct fracture classification and postoperative evaluation in patients with ankle fractures.

DETAILED DESCRIPTION:
History and current related studies Intraarticular fractures and ruptures of ligaments around the joint often occur after ankle injury. Early correct treatment can effectively help joint repair, and reduce the incidence of serious complications. Ankle fractures are one of the common orthopedic fractures. X-ray is a common method for detecting ankle injury, can determine the fracture site, type and extent. However, X-ray is difficult to display ankle fracture, bone fragments, displacement, or ligament injury, so it cannot make accurate fracture classification or formulate treatment programs.

Magnetic resonance imaging (MRI) can clearly show the ankle ligament, tendon, and cartilage injury, is advantageous in the diagnosis of ligament injury after ankle fracture, and can provide accurate imaging information. MRI can provide accurate preoperative assessment of clinical indicators for the rational formulation of treatment programs to reduce complications. The observation of ankle contusion observed by MRI is conducive to analyzing the mechanism of ankle joint injury.

Therefore, X-ray combined with MRI would perfectly verify soft tissue injury after ankle fractures so as to make effective surgical program.

Adverse events Adverse events including incision pain, incision nonunion, ankle pain, peripheral nerve injury of ankle joint, ankle joint inflammation, and soft tissue injury. Severe adverse events are events occurred during clinical trial, including requiring hospitalization, prolonged hospitalization, disability, inability to work, life-threatening, or fatalities. If severe adverse events occur, investigators would report details, including the date of occurrence and measures taken to treat the adverse events, to the principle investigator and the institutional review board within 24 hours.

Data collection, management, analysis and open-access

1. Case report forms with demographic data, disease diagnosis, accompanying diseases, drug allergy history, and adverse events were collected.
2. Data were processed using Epidata software (Epidata Association, Odense, Denmark), collated, and then recorded electronically. All data regarding this trial were preserved by the First Hospital, Hebei Medical University, China.
3. The electronic database was statistically analyzed by a professional statistician who created an outcome analysis report that was submitted to the lead researchers.

ELIGIBILITY:
Inclusion Criteria:

* Ankle fractures patients detected by X-ray
* Highly suspected ankle ligament injury
* History of obvious trauma
* Complete clinical data
* Irrespective of sex and age
* Sign the informed consent

Exclusion Criteria:

* Cardiopulmonary function cannot tolerate anesthesia or surgery
* Open fractures of ankle joint
* Old fracture of the ankle joint

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with excellent effects | at postoperative 3 months
  higher value indicates better repair effect

SECONDARY OUTCOMES:
patients with Lauge-Hansen classification | baseline
  According to the degree of bone and ligament injury, there are supination-external rotation (supination-eversion), pronation-external rotation (pronation-eversion), supination-adduction and pronation-abduction.
X-ray examination | baseline and 3 months postoperatively
  To evaluate the healing degree of fracture
MRI findings | baseline and 3 months postoperatively
  To evaluate ligament repair effects

CONTACTS AND LOCATIONS:
Overall Officials: Guobin Liu, Master, Principal Investigator — The First Affiliated Hospital of Hebei Medical University

IPD SHARING:
Plan to Share IPD: Undecided